CLINICAL TRIAL: NCT06149832
Title: Treatment of Oral Chronic Graft-versus-host Disease With Human Umbilical Cord Mesenchymal Stem Cell Dressing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, ShiCang Yu, director of Stem cell and regenerative medicine, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cGVHD001
Record Dates: First submitted 2023-11-06; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Mesenchymal Stem Cells
Keywords: Oral Chronic Graft-versus-host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs treatment group (Experimental)
  Interventions: Biological: Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSCs) — The patient's mouth (including buccal mucosa, tongue and lip) was applied with MSCs: MSCs (1×10^6/ml) dressing was applied 4 times/day for 2 weeks.

SUMMARY:
Chronic graft-versus-host disease (cGVHD) is a clinicopathological syndrome caused by donor lymphocytes attacking the recipient's organs during the process of reestablishing donor immunity after allogeneic hematopoietic stem cell transplantation (allo-HSCT), with an incidence of about 30%-70%. The clinical manifestations of cGVHD are varied, the course of the disease is prolonged, and the quality of life of patients is affected, and the long-term survival is affected. Among them, oral cGVHD is the most common type, which mainly presents with lichen planus, oral ulcers, mucosal atrophy, erythema and pain. At present, the treatment of oral cGVHD is based on systemic treatment and local hormone-containing gargling solution and local photochemotherapy. The former is easy to be complicated by oral local fungal infection, while the latter has no such equipment in China. Therefore, it is urgent to establish a simple, effective and low-toxicity local treatment for oral cGVHD. Mesenchymal stem cells (MSCs) are one of the most widely used cell products in clinic. The combination of MSCS and hematopoietic stem cells can improve the success rate of transplantation and accelerate hematopoietic reconstruction. The applicant team previously completed a national multi-center clinical study on MSCs prevention of cGVHD, which proved that sequential infusion of MSCs can effectively reduce the incidence of cGVHD, and the mechanism is that MSCs regulate Th1: Th2 balance and promote the differentiation of T cells to Th1 direction. Our previous mechanism study provides an important theoretical basis for MSCs treatment of oral cGVHD. According to the clinical needs and the rich experience of our research group in the field of MSCs clinical research, we plan to use dressing containing MSCs for the local treatment of oral cGVHD, so as to improve the lesion degree of oral cGVHD and improve the quality of life of allo-HSCT patients, and provide clinical experience for reference for the local treatment of MSCs graft-versus-host disease.

ELIGIBILITY:
Inclusion Criteria:

1. No gender limitation, age <65 years old; KPS score >60, estimated survival >3 months.
2. No serious damage to the function of major organs of the whole body.
3. Donor hematopoietic reconstruction was stable (neutrophils >0.5×10^9/L, platelets >20×10^9/L).
4. Stable control of primary blood diseases.
5. Voluntary examination, informed consent.

Exclusion Criteria:

1. Have severe heart, kidney or liver dysfunction.
2. Those combined with other malignant tumors need treatment.
3. There are clinical symptoms of brain dysfunction or severe mental illness and the inability to understand or follow the research protocot4. Patients who cannot be guaranteed to complete the necessary treatment plan and follow-up observation.

5. Patients with severe acute allergic reactions. 6. Clinically uncontrolled active infection. 7. Patients who are participating in other clinical trials. 8. Researchers believe that the subject is not suitable for clinical trials for other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Oral cGVHD improves condition | after 2 weeks of treatment
  Oral cGVHD score

CONTACTS AND LOCATIONS:
Overall Officials: Lei Gao, Study Chair — Army Medical University, China
Locations (1):
- Xinqiao Hospital, Shapingba, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT06149832/Prot_000.pdf